CLINICAL TRIAL: NCT05512091
Title: Characterization of the Pattern of Consumption and Withdrawal Syndrome From Dual Cannabis and Tobacco Use in People With Cannabis Use Disorder Who Initiate Dishabituation Treatment (DuCATA_GAM-CAT)
Brief Title: Characterization of the Pattern of Consumption and Withdrawal Syndrome From Dual Cannabis and Tobacco Use
Acronym: DuCATA_GAMCaT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cristina Martínez Martínez (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); University of Barcelona (Other); Public Health Agency of Barcelona (Other)
Responsible Party: Sponsor-Investigator, Cristina Martínez Martínez, Principal Investigator, Institut Català d'Oncologia
Organization: Institut Català d'Oncologia (Other)
Other Study IDs: DUCATA_GAM-CaT_REF:2020I034
Record Dates: First submitted 2022-05-06; First posted 2022-08-23 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cannabis Dependence; Tobacco Use; Withdrawal Syndrome; Substance Abuse
Keywords: Cannabis; Tobacco; Treatment; Social network
MeSH Terms: conditions — Marijuana Abuse; Tobacco Use; Substance Withdrawal Syndrome; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aims: To characterize the pattern of cannabis and tobacco use and withdrawal symptoms in people who start treatment for cannabis use disorders (exclusive cannabis, concurrent and/or simultaneous with various tobacco products) through an aplication game and considering the type of users. Methodology: Mixed-methods research composed of three studies. Study I: qualitative participatory action study aimed at exploring the experiences and preferences of the cannabis users on the use of apps. This information will be instrumental in the co-design of the app. Study II: prospective longitudinal study aimed to establish consumption patterns and transitions between substances and to validate the scale of cannabis withdrawal symptoms in the Spanish population. Sample size: expected RR=1.20, α =0.05, β= 0.20, losses= 20% (n=282). Study III: qualitative study to explore participants' experiences during the process of quitting cannabis and / or tobacco. Expected results: Characterization and prediction of variables that influence cannabis and tobacco cessation/ reduction and describe withdrawal symptoms according to consumption patterns with aim of improving the design of future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Smokers (at least 1cig./week)
* Undertreatment for Cannabis
* >=18 years-old
* Under clinical follow-up
* Informed consent
* Have a Smartphone

Exclusion Criteria:

* Severe cognitive impairment
* 3-month follow-up not guaranteed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smokers under treatment for cannabis substance abuse from the province of Barcelona in Catalonia (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cannabis use | Change between baseline and 6 weeks follow-up
  Number of participants that use several cannabis products (hashish, marijuana, etc.)
Tobacco use | Change between baseline and 6 weeks follow-up
  Number of participants that use several type of tobacco product/s
Abstinence from cannabis | Change between baseline and 6 weeks follow-up
  If a participant reduces or quits their cannabis use, we will ask for their presence of 16 withdrawal symptoms. Each symptom is scored from 0 (minimum) to 3 (maximum). Higher scores mean a worse outcome.
Abstinence from tobacco | Change between baseline and 6 weeks follow-up
  If a participant reduces or quits their tobacco use, we will ask for their presence of 6 withdrawal symptoms using the Fagerström test. The test has a minimum score of 0 and a maximum of 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Motivation to quit | Baseline
  Using a Likert scale randing from 0 to 10 (0=totally unmotivated and 10= totally motivated)
Psychological assessment | Baseline
  States of change or readiness to quit cannabis and tobacco according to Prochaska and Di Clemente's model (pre-contemplative, contemplative, prepared, action and maintenance.
Self-perceived health status | Baseline
  Will be assessed based on "How would you say your general health is?" (excellent, very good, good, fair, very fair, poor)
Social and cultural factors | Baseline
  Questions related to their social circle/network (friends and colleagues) and social climate overall

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saura J, Enriquez M, Feliu A, Roca X, Mondon S, Barrio P, Andreu M, Segura L, Ballbe M, Fu M, Fernandez E, Martinez C; DuCATA clinical group. Consumption patterns and withdrawal symptoms in dual cannabis-tobacco users in Spain: Cross-sectional study. Addict Behav Rep. 2025 Dec 17;23:100656. doi: 10.1016/j.abrep.2025.100656. eCollection 2026 Jun. PMID 41531671
- [Derived] Saura J, Feliu A, Enriquez-Mestre M, Fu M, Ballbe M, Castellano Y, Pla M, Rosa N, Radeva P, Maestre-Gonzalez E, Cabezas C, Colom J, Suelves JM, Mondon S, Barrio P, Andreu M, Raich A, Bernabeu J, Vilaplana J, Roca Tutusaus X, Guydish J, Fernandez E, Martinez C. Patterns of Use and Withdrawal Syndrome in Dual Cannabis and Tobacco Users (DuCATA_GAM-CAT): Protocol for a Mixed Methods Study. JMIR Res Protoc. 2024 Sep 19;13:e58335. doi: 10.2196/58335. PMID 39298750